CLINICAL TRIAL: NCT07400861
Title: Trial of a New Software Tool for Personalized Minimum and Maximum Pressure Recommendations in New CPAP Users With OSA
Brief Title: Study of Min-Max APAP Recommender Tool
Acronym: SMART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MA011025
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APAP Pressure Match (Experimental): CPAP clinical min-max pressure settings provided by the APAP Pressure Match recommender tool. The tool utilizes machine learning to identify optimal clinical settings for each patient.
  Interventions: Device: CPAP with min-max recommender tool
- Default CPAP settings (Placebo Comparator): Default out-of-box min and max settings for CPAP.
  Interventions: Device: CPAP with default settings

INTERVENTIONS:
Device: CPAP with min-max recommender tool — CPAP where the settings are personalized to each patient, recommended by Pressure Match tool.
  Arms: APAP Pressure Match
Device: CPAP with default settings — CPAP set up on default out-of-box clinical pressure settings.
  Arms: Default CPAP settings

SUMMARY:
Pressure Match (The APAP Min-Max tool) is a software-based clinical decision-support tool, developed using a causal-inference modelling approach based on data from thousands of OSA patients. The model takes as inputs from patient variables (e.g., baseline AHI, gender, weight/BMI, mask interface type), and outputs recommended AutoSet minimum and maximum pressure settings (cmH₂O) tailored for that patient phenotype.

The intended clinical role of the Pressure Match tool is to assist the clinician's choice of AutoSet pressure range when initiating CPAP therapy, with the goal of reducing clinician time/effort in manual titration and follow-up adjustments without compromising safety, efficacy or patient satisfaction.

The purpose of this trial is to test Pressure Match in a clinical trial setting, to demonstrate non-inferiority against standard APAP settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to give written informed consent
* Patients who can read and comprehend English
* Patients who are ≥ 18 years of age
* Patients newly diagnosed with OSA (AHI ≥ 5) and indicated for CPAP therapy.

Exclusion Criteria:

* Patients who have previously used PAP therapy
* Patients who require a bilevel device
* Patients who are or may be pregnant
* Patients with a preexisting lung disease/ condition that would predispose them to pneumothorax (for example: COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection; lung injury
* Patients whose physician has dictated specific therapy settings (e.g. fixed pressure CPAP, or specific AutoSet minimum and/ or maximum settings)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Mean residual AHI | 3 months
  The primary endpoint is comparison of the mean residual AHI of the active group compared with the control group, to demonstrate non-inferiority.
  Apnea-Hypopnea Index (AHI) is defined as the number of obstructive apnea and hypopnea events per hour of sleep. Apneas are episodes of complete cessation of airflow, and hypopneas are episodes of partial reduction in airflow.
  Residual AHI is the AHI calculated from device-recorded data via validated detection algorithms collected while the participant is receiving therapy with the study device. Residual AHI reflects the frequency of obstructive respiratory events that remain during treatment and is used to assess treatment effectiveness.

CONTACTS AND LOCATIONS:
Locations (1):
- West Australian Sleep Disorders Research Institute, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No
IP protected